CLINICAL TRIAL: NCT07281326
Title: A Phase I Study of Evaluating Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of AK138D1 in Advanced Solid Tumors
Brief Title: A Study of AK138D1 in Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK138D1-102
Record Dates: First submitted 2025-09-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Solid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK138D1 (Experimental): AK138D1 will be administered in pre-specified dose levels.
  Interventions: Drug: AK138D1

INTERVENTIONS:
Drug: AK138D1 — Enrolled subjects will receive intravenous infusion (IV) of AK138D1 according to the dosing regimen specified in their cohort.

SUMMARY:
This is a Phase I clinical trial testing the safety and effectiveness of AK138D1in patients with advanced cancer. The study will enroll up to 200 patients with various types of advanced solid tumors who haven't responded to standard treatments. Patients will receive AK138D1 to determine the safest dose and evaluate if the drug can help treat their cancer.

DETAILED DESCRIPTION:
This open-label, dose-escalation and expansion Phase I clinical trial aims to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary anti-tumor activity of AK138D1 in subjects with advanced malignant tumors. The study will test different doses of AK138D1 to find the recommended dose for future studies and assess whether the drug shows signs of effectiveness against cancer. Participants will receive AK138D1 through intravenous infusion and will be closely monitored for side effects and treatment response. The final number of participants enrolled will depend on the safety and effectiveness results observed during the study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must sign the written informed consent form (ICF) voluntarily;
2. At enrollment, aged ≥ 18 to ≤ 75 years, both males and females are eligible;
3. ECOG performance status score of 0 or 1;
4. Has a life expectancy of ≥ 3 months;
5. At least 1 measurable lesion as per RECIST v1.1 that is suitable for repeated accurate measurement.
6. Adequate organ function.

Exclusion Criteria:

1. Prior human epidermal growth factor receptor 3 (HER3) -targeted therapies, including antibodies, antibody-drug conjugates (ADCs), chimeric antigen receptor T-cell immunotherapy (CAR-T), and others;
2. Concomitant participation in another clinical study, unless it is a non-interventional clinical study or the follow-up period of an interventional study;
3. Presence of active central nervous system (CNS) metastases.
4. Live vaccines or attenuated live vaccines administered within 4 weeks prior to the first dose, or planned to be administered during the study; use of inactivated vaccines is allowed;
5. Untreated subjects with active hepatitis B or active hepatitis C;
6. Known active pulmonary tuberculosis (TB); subjects with suspected active TB must undergo appropriate clinical assessment to rule out the presence of active disease;
7. Known active syphilis infection;
8. Subjects with known allergy to any component of any study drug; and with a history of known severe hypersensitivity reactions to other monoclonal antibodies;
9. Other reasons for ineligibility as evaluated by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to approximately 2 years
  Incidence and severity of participants with adverse events
Dose-Limiting Toxicity (DLT) | Up to approximately 2 years
  Occurrence of DLTs and determination fo maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of AK138D1 | Up to approximately 2 years
  AK138D1 serum drug concentrations in subjects at different time points after administration.
Area under the plasma concentration versus time curve (AUC) of AK138D1 | Up to approximately 2 years
  The definite integral of the concentration of AK138D1 in blood plasma as a function of time.
Anti-drug antibodies (ADA) | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies (ADA).
Objective Response Rate (ORR) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , assessed by investigators based on RECIST v1.1.
Disease Control Rate (DCR) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1.
Duration of response (DoR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Duration of response (DoR) assessed according to RECIST v1.1.
Progression Free Survival (PFS) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented disease progression (per RECIST v1.1 criteria) assessed by investigators or death due to any cause, whichever occurs first.
Time to response (TTR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  Time to response (TTR) is defined as the time to response based on RECIST v1.1.
Overall Survival (OS) | Up to approximately 2 years
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wenting Li, MD, Study Director — Akeso
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No